CLINICAL TRIAL: NCT02772211
Title: D-cycloserine for Relapse Prevention Following Intravenous Ketamine in Treatment-resistant Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Teva Pharmaceuticals USA (Industry); Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Revital Amiaz, Doctor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2853-15-SMC
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-cycloserine (Experimental): Participants in this group would receive 6 infusions of ketamine. Participants who demonstrate symptoms reduction following ketamine infusions would receive oral D-cycloserine, titrated slowly up to 1000mg/d over the next 8 weeks.
  Interventions: Drug: Ketamine; Drug: D-cycloserine
- Placebo (Placebo Comparator): Participants in this group would receive 6 infusions of ketamine. Participants who demonstrate symptoms reduction following ketamine infusions would receive oral Placebo pills, titrated slowly up to 1000mg/d over the next 8 weeks.
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Patients will undergo 6 ketamine infusions within a 3-week period. Intravenous ketamine will be administrated by a senior anesthesiologist and under the supervision of a senior psychiatrist hence ensuring patient safety. The procedure will be explained in detail to each patient, and written consent will be obtained.
  After a psychiatric and medical evaluation by a senior psychiatrist and a senior anesthesiologist, patients will be given ketamine infusion added on to their antidepressant therapy. A slow ketamine infusion of 0.5mg/kg over 40 minutes will be given to the patients. Patients will be monitored by the experienced staff which includes a senior anesthesiologist and a nurse as well as a psychiatrist who will be available nearby. All patients will be monitored continuously for heart rate and rhythm and oxygen saturation, and blood pressure will be measured at 10 minutes intervals.
Drug: D-cycloserine — Following completion of Ketamine infusions. patients in the experimental group will start receiving D-cycloserine pills titrated slowly up to 1000mg/d over the next 8 weeks [2] in the following manner:
  1. Week 4: Days 22-24 - 250mg/d, one pill per day Well-being assessment and adverse effect evaluation before drug elevation.
  2. Mid-week 4 to end of week 6: Days 25-42 - 500mg/d, two pills per day
  3. Week 7: Day 43-49 - 750mg/d, three pills per day
  4. Weeks 8-11: Days 50-77 - 1000mg/d four pills per day
  Other Names: D-cycloserine, Cycloserine, DCS
  Arms: D-cycloserine
Drug: Placebo — Following completion of Ketamine infusions. patients in the experimental group will start receiving placebo titrated slowly up to 1000mg/d over the next 8 weeks [2] in the following manner:
  1. Week 4: Days 22-24 - 250mg/d, one pill per day Well-being assessment and adverse effect evaluation before drug elevation.
  2. Mid-week 4 to end of week 6: Days 25-42 - 500mg/d, two pills per day
  3. Week 7: Day 43-49 - 750mg/d, three pills per day
  4. Weeks 8-11: Days 50-77 - 1000mg/d four pills per day
  Arms: Placebo

SUMMARY:
This is a two-stage experiment; the first stage is an open label trial in which participants receive six intravenous (IV) treatments of ketamine. The second stage includes participants that responded to ketamine (i.e. reduction of 25% in their symptoms of depression, as measured by the Montgomery Asberg Depression Scale MADRS). The second stage is a double-blind, controlled clinical trial of D-cycloserine (DCS) vs. placebo, as maintenance treatment in patients who responded to ketamine treatment. The aim of the study is to determine whether 8 weeks of DCS maintenance therapy will prevent relapse of depressive symptoms following ketamine infusions

DETAILED DESCRIPTION:
Background MDD is one of the leading causes of disability worldwide [5]. A substantial proportion of patients do not achieve adequate remission despite multiple antidepressant trials and augmentation strategies. TRD is defined as an insufficient response to at least two adequate antidepressant trials. Many of these patients are referred to somatic treatment; e.g. electroconvulsive therapy (ECT), repetitive Transcranial Magnetic Stimulation (rTMS) and Vagal Nerve Stimulation (VNS), all of which can cause side effects, and are not always efficacious.

Ketamine has been safely used for decades for the induction and maintenance of anesthesia and more recently for chronic pain. Ketamine is a noncompetitive, high-affinity antagonist of the NMDA type glutamate receptor, with additional effects on dopamine and μ-opioid receptors. During the last decade, 4 meta analyses summarizing over 22 controlled trials have been published, showing the rapid and impressive effect of ketamine in TRD patients [6-8]. These trials show that a single slow IV ketamine sub-anesthetic dose (0.5 mg/kg) over 40 minutes dramatically improves depressive symptoms. Across studies, a clinically significant antidepressant response was maintained for up to 72 hours in approximately half of the patients; only a minority had relapsed within the first two weeks post-ketamine infusion [9, 10]. aan het Rot et al. [11] showed that repeated IV ketamine infusions prolong the duration of improvement.

D-cycloserine (seromycin) is a broad spectrum antibiotic, in use for over thirty years in the treatment of tuberculosis, DCS functions as a partial agonist at the NMDA-R glycine site, with agonist effects predominating at low dose and antagonist effects at high dose. Low DCS dosages, such as 50-500 mg/d have been implemented in anxiety patients for memory and learning enhancement. Beneficial antidepressant effects have been reported when higher dosages (500-1000 mg/day) were used [3]. DCS regimens in TRD patients suggest that high dose DCS may indeed be beneficial in the treatment of MDD. However, a previous study using a lower dosage (250mg/d) did not show significant difference over placebo [3]. The antidepressant effects of DCS seem to derive from its ability to inhibit NMDA-R function, similarly to ketamine. One recent study demonstrated a beneficial effect of DCS after ketamine infusion in bipolar depression patients [12]. Due to the potential neurotoxicity of ketamine in prolonged administration. Other NMDA antagonist should follow ketamine infusion [13]. Therefore we reason that DCS post-ketamine administration will considerably reduce relapse in TRD patients when compared to placebo.

Study Design

1. Patients will undergo 6 ketamine infusions within a 3-week period.

   Intravenous ketamine will be administrated by a senior anesthesiologist and under the supervision of a senior psychiatrist hence ensuring patient safety. We believe that sub-anesthetic ketamine infusion will be safer and will cause fewer side effects than ECT. The procedure will be explained in detail to each patient, and written consent will be obtained.

   After a psychiatric and medical evaluation by a senior psychiatrist and a senior anesthesiologist, patients will be given ketamine infusion added on to their antidepressant therapy. A slow ketamine infusion of 0.5mg/kg over 40 minutes will be given to the patients. Patients will be monitored by the experienced staff which includes a senior anesthesiologist and a nurse as well as a psychiatrist who will be available nearby. All patients will be monitored continuously for heart rate and rhythm and oxygen saturation, and blood pressure will be measured at 10 minutes intervals. Heart rate variability will be measured and analyzed after ketamine treatment. Measurements will be performed during the ketamine infusion at baseline, after 3 and 6 treatments. Depressive symptoms will be measured using Montgomery Asberg Depression Scale (MADRS). In addition Clinical Global Severity Scale (CGI-S) and Clinical Global Improvement (CGI-I) will be performed 2 hours after treatment. In many cases, patients with depression also suffer from alexithymia: inappropriate identification of emotions. Alexithymia will be measured at baseline after 3 and 6 treatments. Ketamine infusion will be stopped in cases of a 20% or above increase in blood pressure or in heart rate over baseline values and/ or an acute dissociative state.

   Patients will be discharged to their homes at least three hours from end of infusion. Due to the potential effect of ketamine each patient will need to be escorted to and from the hospital by a family member or a friend.
2. For patients who will meet response criteria (MADRS≥25%) after 6 ketamine infusions, ketamine administration (weeks 1-3: days 1-21) will be stopped and patients will start receiving DCS or placebo titrated slowly up to 1000mg/d over the next 8 weeks [2] in the following manner:

   1. Week 4: Days 22-24 - 250mg/d, one pill per day Well-being assessment and adverse effect evaluation before drug elevation.
   2. Mid-week 4 to end of week 6: Days 25-42 - 500mg/d, two pills per day
   3. Week 7: Day 43-49 - 750mg/d, three pills per day
   4. Weeks 8-11: Days 50-77 - 1000mg/d four pills per day
3. Pyridoxine 200-300mg/d will be prescribed for all patients at the beginning of the study.
4. Patients who did not improve after 6 ketamine treatments will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 meeting DSM-V criteria for moderate-severe depression (MADRS≥25), who did not respond to two adequate antidepressant courses of treatment. Subjects will be required to continue on a stable dose of any psychotropic medication they are taking, for 8 weeks prior to ketamine infusion. Participants who respond to ketamine (reduction of 25% in symptoms) would be invited to participate in a second stage of the experiment, in which participants would consume DCS for 8 weeks (weeks 4-11).

Exclusion Criteria:

* Patients will be excluded if they have current or history of psychotic or dissociative symptoms, or severe personality disorder with psychosis or dissociative symptoms. Additional exclusion criteria will be a lifetime history of psychotic mania, a substance abuse or use of alcohol. Medical exclusion criteria will include - uncontrolled elevated blood pressure, non-sinus rhythm, unstable ischemic heart disease, uncorrected hyper thyroidism, and for women, pregnancy or the initiation of female hormonal treatment <3 months. Before ketamine treatment women of childbearing age will be required to use a medical accepted contraceptive or abstain from sexual activity. In addition patients will be excluded if they suffer from chronic renal failure, epilepsy, organic brain disorder or neurological or an unstable medical condition. Due to neurotoxicity and convulsions, patients will be prohibited to consume alcohol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Scale (MADRS) | screening criteria, after third ketamine infusions
  A diagnostic questionnaire, measuring the severity of depressive episodes.

OTHER OUTCOMES:
Hamilton depression Rating Scale | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
  A diagnostic questionnaire, measuring the severity of depressive episodes.
Clinical Global Severity Scale | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
  A questionnaire, measuring the current global state of a person
Clinical Global Improvement | after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
  A questionnaire, measuring the improvement in clinical symptoms
Hamilton Anxiety Scale | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
Toronto Alexithymia Scale | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
N-Back test | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
  computerized tasks featuring neutral stimuli
Verbal Fluency test | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
  computerized tasks featuring neutral stimuli
Stop signal test | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
  computerized tasks featuring neutral stimuli
ANTI | Up to ten days pre first ketamine administration, after third ketamine infusion, after sixth ketamine infusion, week 7, week 11, 2 months after study completion
  computerized tasks featuring neutral stimuli

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatry Clinic - Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No